CLINICAL TRIAL: NCT00923039
Title: The Early Origins of Cardiovascular Disease : the Consequence of Growth Restriction During Foetal Life and Infancy on Cardiovascular Structure and Function in Adulthood
Brief Title: The Early Origins of Cardiovascular Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Danone Institute International (Other)
Responsible Party: Dardaine /General representative, Danone Institute International
Other Study IDs: NU 304
Record Dates: First submitted 2009-06-17; First posted 2009-06-18 (Estimated); Last update posted 2009-06-18 (Estimated); Status verified 2009-06

CONDITIONS: Cardiovascular Disease
Keywords: The early origin of cardiovascular disease
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

GROUPS / COHORTS (1):
- Exposed/ Not exposed

SUMMARY:
Small body size at birth, slow weight gain during infancy and increase in body mass index after 2 years are independent risk factors for cardiovascular disease and the metabolic syndrome. There is a large gap in our understanding of how early growth affects the cardiovascular system. Possible mechanisms include alterations in body composition, in cardiac structure, in vascular function, in renal function and epigenetic processes.

The Objective is to determine how size at birth and growth during infancy and childhood affect: body composition, cardiac structure and function, vascular and endothelial function, renal function, metabolic status and transcriptional and epigenetic characteristics.

ELIGIBILITY:
Inclusion Criteria:

* Male and female volunteers students aged between 18-25 years old
* Having growth records

Exclusion Criteria:

* If young women subject without contraception,or pregnant

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: 200 Young adult students will be recruited at the Preventive Medicine Centre at Université de la Méditerranée during their annual routine medical examination
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2009-06

PRIMARY OUTCOMES:
To determine how size at birth and growth during infancy and childhood affect: body composition, cardiac structure and function, vascular and endothelial function, renal function, metabolic status and transcriptional and epigenetic characteristics | 3 years

CONTACTS AND LOCATIONS:
Locations (1):
- CIC-UPCET Hopital de la Timone Bat F, Marseille, France